CLINICAL TRIAL: NCT04308317
Title: Clinical Study of Tetrandrine Tablets Adjuvant Treatment With COVID-19
Brief Title: Tetrandrine Tablets Used in the Treatment of COVID-19
Acronym: TT-NPC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-NPC
Record Dates: First submitted 2020-03-04; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Corona Virus Disease 2019,COVID-19
Keywords: COVID-19; Tetrandrine
MeSH Terms: conditions — COVID-19 | interventions — tetrandrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetrandrine Cohort (Experimental): After the subjects were enrolled, they were given "Tetrandrine 60mg QD" for a course of 1 week(Take 6 days, stop using for 1 day)
  Interventions: Drug: Tetrandrine
- Control Cohort (No Intervention): Treatment according to standard protocols without intervention

INTERVENTIONS:
Drug: Tetrandrine — Tetrandrine 60mg QD for 1week
  Other Names: tetrandrine tablets
  Arms: Tetrandrine Cohort

SUMMARY:
The study is expected to treat patients with mild and severe neo-coronary pneumonia through standard treatment regimens in combination with tetrandrine tablets, thereby reducing the clinical progress of some patients, improving prognosis, reducing the incidence of pulmonary fibrosis during rehabilitation, and improving patients' quality of life.

DETAILED DESCRIPTION:
Since December 2019, a number of cases of pneumonia infected with the new coronavirus have been found in wuhan, hubei province.Has now become a global epidemic of crisis.

After recent frontline anti-epidemic experience, the diagnostic and treatment specifications for new coronary pneumonia have been updated several times. In the latest country, "Specifications for the Diagnosis and Treatment of New Types of Coronary Pneumonia (Trial Version 6)", the traditional Chinese medicines have again emphasized For the treatment of patients, traditional Chinese medicine preparations such as Xuebijing and Qingfei Paidu Decoction have been recommended, but the introduction of anti-fibrosis related drugs is still lacking.Tetrandrine is a traditional Chinese medicine. Previous research has shown that it is an antagonist of calmodulin, has anti-tumor, anti-inflammatory effects, and can effectively inhibit fibroblasts, thereby inhibiting pulmonary fibrosis.The study is expected to treat patients with mild and severe neo-coronary pneumonia through standard treatment regimens in combination with tetrandrine tablets, thereby reducing the clinical progress of some patients, improving prognosis, reducing the incidence of pulmonary fibrosis during rehabilitation, and improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild and severe cases who have been diagnosed with new coronavirus pneumonia according to the "Pneumonitis Diagnosis and Treatment -
* Plan for New Coronavirus Infection"
* Age 18 to 75 years;
* Sign the informed consent voluntarily.

Exclusion Criteria:

* With active tuberculosis, idiopathic pulmonary fibrosis, bronchial asthma, bronchiectasis, pulmonary embolism, patients with chronic respiratory failure or other severe respiratory disease;
* According to the "pneumonia diagnosis and treatment program for new coronavirus infection" (trial version 6), critically ill patients
* With severe patients with disease of heart head blood-vessel, malignant arrhythmia, unstable angina, acute myocardial infarction and death, cardiac function level 3 and above, stroke, cerebral hemorrhage, etc.);
* With severe liver and kidney diseases (severe liver disease refers to cirrhosis, portal hypertension and varices bleeding, severe kidney disease including dialysis, kidney transplantation);
* Pregnant and lactating women;
* Severe cognitive and mental disorders;
* Clinical investigators who were participating in other interventions within 1 month prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 12 weeks
  Death event

SECONDARY OUTCOMES:
body temperature | 2 weeks
  inflammatory indicator

CONTACTS AND LOCATIONS:
Locations (1):
- Tetrandrine Tablets, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No